CLINICAL TRIAL: NCT05238532
Title: A Multi-center, Open-label Dose-escalation and Dose-finding Phase I Clinical Trial to Evaluate the Safety, Tolerability and Efficacy of CT303 in Patients With Acute Respiratory Distress Syndrome
Brief Title: Clinical Trial to Evaluate the Safety, Tolerability and Efficacy of CT303 in Patients With ARDS
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulties in recruiting Subjects
Sponsor: GC Cell Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT303B101
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): CT303
  Interventions: Genetic: CT303

INTERVENTIONS:
Genetic: CT303 — Once a time, intravenous injection
  * CT303 Starting Dose : 1.0*10^6 cells/kg
  * CT303 Increasing Quantity Dose : 2.0*10^6 cells/kg

SUMMARY:
Evaluate the safety, tolerability, efficacy and pharmacodynamics&pharmacokinetic properties of CT303 in patients with ARDS.

DETAILED DESCRIPTION:
This study is a multi-center, open-label, dose-escalation and dose-finding phase 1 clinical trial.

The primary purpose is to evaluate the safety and tolerability of CT303 and the Secondary purpose is to evaluate the efficacy of CT303 in patients with ARDS. And the exploratory purpose is to evaluate pharmacodynamics properties pharmacokinetic properties of CT303 in patients with ARDS.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 19 years old
* Patients who meet the ARDS criteria according to the Berline definition

  1. within 1 week of a known clinical insult or new or worsening respiratory symtoms
  2. Bilateral opacities not fully explained by effusions, loar/lung collapse, or nodules
  3. Respiratory failure not fully explained by cardiac failure or fluid overload
  4. oxygenation corresponding to mild, moderate, severe
* Patients requiring positive pressure ventilation using an endotracheal tube
* Patients or legal representative signed Informed consent form

Exclusion Criteria:

* Greater than 96 hours since first meeting ARDS criteria
* Patients who was previously administered mesenchymal stem cell therapy products or other cell therapy products
* Patients with the following medical history or comorbid condition

  1. medical history

     1. Patients who had an organ transplant or bone-marrow transplantation
     2. Patients who had a pneumonectomy
     3. a maligant tumor within 5 years
     4. a deep vein thrombosis or pulmonary embolism with in 6 months
     5. a trauma within 7 days
  2. comorbid condition

     1. Patients with AST or ALT exceeding 5 times the upper limit of the normal range
     2. eGFR ≤ 29mL/min or Patients requiring continuous renal replacement therapy
     3. severe chronic respiratory disease
     4. WHO functional assessment class III/IV pulmonary hypertension
     5. Severe cardiac insufficiency
     6. QTc > 480msec
     7. chronic underlying diseases
* viral hepatitis type B or type C, or positive HIV test
* Patients using extracorporeal life support devices or high-frequency oscillatory ventilation
* Moribund patients expected to die within 48 hours
* Patients who refuse or are likely to refuse life-sustaining treatment
* Fertile women or men who disagree a continence and a contraception
* Patients with a history of hypersensitivity reaction
* Patients participating in clinical trials within 4 weeks
* Patients determined by the investigator to be inappropriate to participate in this clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Adverse Drug Reaction incidence rate | Day 0 to Day 28
  Evaluate safety through the incidence rate of adverse drug reactions corresponding to criteria for stopping the dose increasing.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Jae Cho, MD, MPH, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (3):
- South Korea (3):
  - Seoul national university hospital, Seoul
  - Seoul national university boramae medical center, Seoul
  - Seoul National University Bundang Hospital, Seoul